CLINICAL TRIAL: NCT03595943
Title: A Low Glycemic Index Diet for Prevention of Glucose Intolerance During Bed Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17-176
Record Dates: First submitted 2018-06-27; First posted 2018-07-23 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycemic index diet (Experimental): Low glycemic index pulse-based diet (i.e. beans, peas, lentils, chickpeas)
  Interventions: Dietary Supplement: Low glycemic index, pulse-based diet
- Regular hospital diet (Active Comparator): Moderate glycemic index diet based on hospital menus
  Interventions: Dietary Supplement: Moderate glycemic index hospital diet

INTERVENTIONS:
Dietary Supplement: Low glycemic index, pulse-based diet — Diet that includes pulses (i.e. meals that contain chickpeas, lentils, beans, or peas)
  Arms: Low glycemic index diet
Dietary Supplement: Moderate glycemic index hospital diet — Diet that is derived from a regular hospital menu for patients
  Arms: Regular hospital diet

SUMMARY:
Recovery from surgery, injury or illness might require periods of bed rest in-hospital or at home. Bed rest may be needed for recovery but also has negative consequences. Prolonged bed rest reduces the ability of muscle to take up sugar from the blood, and increases blood levels of sugar and fat which may actually delay recovery. Bone starts breaking down when there is very little skeletal stimulation or 'stress' that typically occurs with walking. Bed rest stiffens arteries which may increase blood pressure. Different diets may influence the extent of harmful effects to muscle, bone and arteries during bed rest. This study compares a diet with increased plant sources (i.e. lentils, chickpeas, beans and peas) to a typical hospital diet (mostly animal sources and foods high in refined sugar) on blood, arteries, muscle and bone during bed rest. The investigators will test six healthy adults before, during and after two periods of 4-day bed rest, one when they eat a typical hospital diet, one with a diet containing more plant sources. The investigators will learn more about the effects of diet during bed rest and be able to make recommendations about diets to help ensure healthy recovery for individuals requiring bed rest.

DETAILED DESCRIPTION:
Many medical conditions and interventions require periods of bed rest in order to maximize recovery and restore optimal physical function. Unfortunately, muscle becomes glucose intolerant, bone starts to break down, and arteries become stiffer during sustained periods of chronic inactivity, such as bed rest. Elevation of blood glucose during hospital stays results in increased morbidity, mortality, length of stay and costs. Components of the typical Western diet (refined carbohydrates and protein from animal sources common in hospital foods) induce glucose intolerance, bone catabolism, and arterial stiffening; plant-based proteins may not have the same negative impact. Pulses (i.e. low fat legumes: lentils, chickpeas, beans, peas) contain carbohydrate with a low glycemic index, and do not substantially increase blood glucose levels. At the same time, they are high in protein, but do not contain the same sulphur-containing amino acid profile as animal proteins that induce bone resorption. Pulses are, therefore, a potential 'super food' to mitigate many of the negative impacts associated with required bed rest following medical illness.

The study purpose is to determine the effects of a pulse-based diet compared to a Western diet of typical hospital foods on glucose tolerance, bone catabolism, and arterial stiffening during bed rest. The investigators hypothesize that a pulse-based diet will be superior to a typical Western diet for preventing glucose intolerance, bone catabolism, and arterial stiffening during sustained bed rest.

Six healthy adults will take part in a cross-over study where they will be randomized to four days of bed rest while on a pulse-based or Western diet, have a one month wash-out and then cross-over before another four days of bed rest with the other diet. Immediately before and after bed rest (i.e. the first morning after the last night of bed rest), oral glucose tolerance tests will be conducted to assess glucose tolerance and insulin sensitivity (i.e. markers used to assess diabetes risk). At the same time points, fasting blood samples will be collected for lipid assessments. Urine will be collected for assessment of bone catabolism (via measures of N-telopeptides: a by-product of collagen from bone which appears in the urine when bone is breaking down). Blood pressure will be evaluated every two hours during bed rest days from 9am to 9pm. Arterial stiffness (measured by the gold-standard technique of pulse wave velocity using applanation tonometry) and beat-by-beat blood pressure will be used to assess blood vessel function before and after four days of bed rest.

This study will inform improved hospital diets and nutritional habits of patients to prevent or offset negative health implications during periods of bed rest that may be required either in-hospital, long-term care or at home as part of standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Diabetic
* Vegetarian
* Food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve | Change from baseline to 4 days
  glucose area under the curve from 2-hour oral glucose tolerance test

SECONDARY OUTCOMES:
Insulin area under the curve | Change from baseline to 4 days
  Insulin area under the curve from 2-hour oral glucose tolerance test
Fasting glucose | Change from baseline to 4 days
  Fasting glucose from serum
Fasting insulin | Change from baseline to 4 days
  Fasting Insulin from serum
Fasting cholesterol | Change from baseline to 4 days
  Fasting cholesterol from serum
Fasting LDL-cholesterol | Change from baseline to 4 days
  Fasting LDL-cholesterol from serum
Fasting triglycerides | Change from baseline to 4 days
  Fasting triglycerides from serum
Fasting HDL-cholesterol | Change from baseline to 4 days
  Fasting HDL-cholesterol from serum
Bone resorption | Change from baseline to 4 days
  Urinary n-telopeptides
Lean tissue mass | Change from baseline to 4 days
  Lean tissue mass from dual energy X-ray absorptiometry scans
Fat mass | Change from baseline to 4 days
  Fat mass from dual energy X-ray absorptiometry scans
Systolic Blood pressure | Change from baseline to 1, 2, 3, and 4 days
  Beat-by-beat blood pressure measurement
Arterial stiffness | Change from baseline to 1, 2, 3, and 4 days
  Arterial stiffness assessed by tonometry
Diastolic blood pressure | Change from baseline to 1, 2, 3, and 4 days
  Beat-by-beat blood pressure measurement

CONTACTS AND LOCATIONS:
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan (SK), Canada

IPD SHARING:
Plan to Share IPD: No